CLINICAL TRIAL: NCT00429143
Title: A Two Step Approach To Allogeneic Hematopoietic Stem Cell Transplantation for Hematologic Malignancies From HLA Partially-Matched Related Donors
Brief Title: A Two-Step Approach to Bone Marrow Transplant Using Cells From A Partially-Matched Relative
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06U.20; 2005-84 (Other: CCRRC); JT 1157 (Other: JeffTrial Number)
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Malignancies
Keywords: Hematologic Malignancies; Two Step Approach; Haploidentical Transplant
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Whole-Body Irradiation; Radiotherapy; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical Allogeneic Transplantation (Experimental): Patients undergoing hematopoietic stem cell transplant from a partially matched related donor
  Interventions: Radiation: Total Body Irradiation (TBI); Biological: Donor Lymphocyte Infusion (DLI); Drug: Cyclophosphamide (CY); Drug: Tacrolimus; Drug: Mycophenolate Mofetil (MMF); Biological: Hematopoietic Stem Cell Transplant (HSCT)

INTERVENTIONS:
Radiation: Total Body Irradiation (TBI) — TBI twice daily days 6-9 prior to transplant (HSCT)
  Other Names: TBI; radiotherapy
Biological: Donor Lymphocyte Infusion (DLI) — DLI given 6 days prior to transplant (HSCT).
  Other Names: DLI; T cell infusion
Drug: Cyclophosphamide (CY) — Cyclophosphamide given once daily at 60 mg/kg on days 2 and 3 prior to transplant (HSCT).
  Other Names: CY; Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Tacrolimus — Tacrolimus given one day prior to transplant (HSCT).
  Other Names: FK-506; fujimycin; Prograf; Advagraf; Protopic
Drug: Mycophenolate Mofetil (MMF) — MMF given one day prior to transplant (HSCT).
  Other Names: MMF; CellCept; Myfortic
Biological: Hematopoietic Stem Cell Transplant (HSCT) — CD34+ selected Hematopoietic Stem Cell Transplant (HSCT) is performed. This is the day of transplantation.
  Other Names: HSCT; stem cell transplant

SUMMARY:
The purpose of this study is to develop a way of treating patients who do not have a completely matched family donor or a readily available unrelated donor with bone marrow transplant by using a partially-matched family donor. Patients receiving this type of transplant will receive chemotherapy and/or radiation to treat their disease. They will also receive their donor's cells in 2 parts. During the first part, the donor's lymphocytes will be exposed to one of the chemotherapy agents to help the patient become tolerant to the lymphocytes. In the second part of the transplant, the patient will receive their donor's stem cells to help recover their peripheral blood counts and establish long-term engraftment. The hypothesis of this study is that in partially-matched allogeneic transplant, there is a defined number of donor T-cells that can be treated and given to the recipient to avoid post-transplant infection without causing severe graft-versus-host disease.

DETAILED DESCRIPTION:
Haploidentical hematopoietic stem cell transplant is a life-saving therapy for patients who are without well matched donors. This type of therapy has been associated with poor outcomes in the past due to complications such as infection. The Jefferson 2 Step approach was designed to allow the infusion of an exact dose of tolerized lymphocytes in haploidentical transplant in order to allow for immune reconstitution post transplant to avoid infectious complications while still having acceptable rates of GVHD. In this approach, patients with high-risk hematological malignancies undergo 8 fractions of TBI (12 Gy) followed by an exact dose of donor lymphocytes. The phase I portion of the study determined the optimal dose of lymphocytes. Two days after receiving the donor lymphocytes, the patients receive 2 daily doses of cyclophosphamide. One day after receiving cyclophosphamide, the patients receive stem cell from their donor. Tacrolimus and mycophenylate mofetil are used as GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematologic or oncologic diagnosis in which allogeneic HSCT is thought to be beneficial, and in whom front-line therapy has already been applied.
2. Patients must have a related donor who is either a one, two or three out of six antigen mismatch at the HLA-A;B;DR loci.
3. Patients without a well-matched unrelated donor or those who have a disease status that precludes a wait for an identified unrelated donor.
4. Patients must adequate organ function:

   * LVEF of >45%
   * FVC or FEV1 >45% of predicted
   * Adequate liver function as defined by a serum bilirubin <1.8, AST or ALT < 2.5X upper limit of normal
   * Serum creatinine < 2.0 mg/dl or creatinine clearance of > 40 ml/min
5. Performance status > 60% (Karnofsky)
6. Patients must be willing to use contraception if they have childbearing potential
7. Able to give informed consent

Exclusion Criteria:

1. An eligible HLA-identical sibling donor.
2. Performance status < 60% (Karnosfsky)
3. HIV positive
4. Active involvement of the central nervous system with malignancy
5. Psychiatric disorder that would preclude patients from signing an informed consent
6. Pregnancy
7. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Grosso D, Carabasi M, Filicko-O'Hara J, Kasner M, Wagner JL, Colombe B, Cornett Farley P, O'Hara W, Flomenberg P, Werner-Wasik M, Brunner J, Mookerjee B, Hyslop T, Weiss M, Flomenberg N. A 2-step approach to myeloablative haploidentical stem cell transplantation: a phase 1/2 trial performed with optimized T-cell dosing. Blood. 2011 Oct 27;118(17):4732-9. doi: 10.1182/blood-2011-07-365338. Epub 2011 Aug 25. PMID 21868572
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to Thomas Jefferson University with hematological malignancies requiring hematopoeitic stem cell transplantation without matched related donors. Opened January, 2006 through August, 2009
Period: Overall Study
Arm/Group | Haploidentical Allogeneic Transplantation
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Haploidentical Allogeneic Transplantation
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Participants
Description: To determine overall survival at 6 months post-transplant.
Time Frame: 6 months
Population: 27 Patients undergoing haploidentical transplant at Thomas Jefferson University
Measure: Number; unit: participants
Arm/Group | Haploidentical Allogeneic Transplantation
Number analyzed (Participants) | 27
participants | 13

2. Primary Outcome: Optimal Dose of CD3+ Donor Lymphocytes (T-cells) for Consistent Engraftment Without GVHD
Description: To determine the optimal dose of CD3+ donor lymphocytes required for consistent engraftment without the development of grade III/IV GVHD.
  Measured as CD3+ donor lymphocytes given as n x 10^8/kg.
  "n" was found to be 2 and was found to be the optimal dose and was the only dose given.
Time Frame: 6 months
Population: Two patients died prior to expected day of engraftment
Measure: Number; unit: lymphocytes x 10^8/kg
Arm/Group | Haploidentical Allogeneic Transplantation
Number analyzed (Participants) | 25
lymphocytes x 10^8/kg | 2

3. Secondary Outcome: Engraftment Rates
Description: To assess hematopoietic engraftment rates.
Time Frame: 6 months
Population: Two patients died prior to expected engraftment day
Measure: Number; unit: participants
Arm/Group | Haploidentical Allogeneic Transplantation
Number analyzed (Participants) | 25
participants | 23

4. Secondary Outcome: Lymphoid Recovery
Description: To assess the pace of lymphoid recovery in this patient population.
Time Frame: 6 months
Population: Two patients did not engraft, two patients died prior to expected day of engraftment
Measure: Number; unit: participants
Arm/Group | Haploidentical Allogeneic Transplantation
Number analyzed (Participants) | 23
participants | 23

5. Secondary Outcome: Incidence of Grades III-IV GVHD
Description: To determine the incidence and severity of GVHD in these patients using a combination of cyclophosphamide, tacrolimus and mycophenolate mofetil (MMF) as GVHD prophylaxis.'
  Severity was graded using CTCAE 3.0 (1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death)
Time Frame: 6 months
Population: Two patients died prior to expected engraftment. Two patients who rejected were retransplanted and were evaluable for GVHD.
Measure: Number; unit: participants
Arm/Group | Haploidentical Allogeneic Transplantation
Number analyzed (Participants) | 25
participants | 2

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Haploidentical Allogeneic Transplantation
Serious Adverse Events (participants affected / at risk) | 23/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Allogeneic Transplantation (N=27)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 (1)
Death - Disease progression NOS (General disorders) | 5 (5)
Liver dysfunction/failure (Hepatobiliary disorders) | 1 (1) — Hepatic failure
Death - Multi-organ failure (General disorders) | 3 (3)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 8 (9)
Infection - Other (Infections and infestations) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 (1)
Constitutional Symptoms - Other (General disorders) | 1 (1)
Death - Death NOS (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Allogeneic Transplantation (N=27)
Mucositis/stomatitis (Gastrointestinal disorders) | 23 (23)
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 (2)
Bilirubin (Metabolism and nutrition disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Limitations of the trial include small sample size and single institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No